CLINICAL TRIAL: NCT05421767
Title: National Tawan University Hospital
Brief Title: Renal Nerve Stimulation in Uncontrolled Hypertensive Patients Undergoing Renal Denervation
Acronym: RND
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201902040RINC
Record Dates: First submitted 2020-04-24; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-04

CONDITIONS: Hypertension
Keywords: renal nerve stimulation; renal nerve denervation; Sympathetic nerve activity
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: RNS checked RDN
Masking Description: RNS guided RDN
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low RNS-induced SBP change group (Active Comparator): 25 patients with the RNS-induced systolic BP change <20mmHg immediately after RDN
  Interventions: Procedure: nerve stimulation guided renal denervation procedure
- High RNS-induced SBP change group (Placebo Comparator): 8 patients with the RNS-induced systolic BP change >20mmHg immediately after RDN
  Interventions: Procedure: nerve stimulation guided renal denervation procedure
- intensive RDN group (Experimental): 17 patients with the initial RNS-induced systolic BP change >20mmHg immediately after RDN, received intensive RDN therapy and let the second RNS-induced systolic BP change < 20mmHg
  Interventions: Procedure: nerve stimulation guided renal denervation procedure

INTERVENTIONS:
Procedure: nerve stimulation guided renal denervation procedure — RNS-in
  Other Names: RNS-guided RDN

SUMMARY:
Study design: Investigator initiated, single center The study is aimed

1) To investigate the blood pressure (BP) change to renal nerve stimulation(RNS), and subsequently perform a renal denervation(RDN) procedure

1) to verify the cutoff value (RNS-induced systolic BP change <20 mmHg in post-RDN patients) could be a useful clinical endpoint in RDN therapy, and test the hypothesis that intense RDN could improve the efficacy of RDN.

DETAILED DESCRIPTION:
Hypertension has become a global public health concern and associated with considerable risk of cardiovascular, cerebrovascular and kidney diseases. Although pharmacological blood pressure (BP) control can reduce these risks, BP control rates remain suboptimal. Resistant hypertension affects 10% to 15% of patients with hypertension and adequate BP control is associated with better clinical outcome of resistant hypertension. Percutaneous renal denervation system (RDN) is designed to disrupt renal afferent and efferent sympathetic nerves to modulate central sympathetic outflow and renal physiology, achieving sustained BP reduction. Although the randomized, sham-controlled trial, SYMPLICITY HTN-3 in 2014, failed to prove the effectiveness of RDN in reducing BP compared to sham procedure, three carefully designed, randomized sham-controlled RDN trials (SPYRAL HTN-OFF MED, SPYRAL HTN-ON MED, and RADIANCE-HTN SOLO), all of which showed similar and clinically meaningful BP reductions without serious adverse events. RDN, therefore, has been approved and well utilized in clinical practice to treat resistant hypertension. However,15-30% of the patients are non-responders. The reason for this is unknown. Experimental data show that renal nerve stimulation (RNS) may serve as a functional endpoint to assess completeness of the RDN procedure. Our preliminary observation study showed low RNS-induced SBP change in post-RDN patients were associated with better BP lowering response.

Our study objectives are

1) to investigate the BP change to RNS, and subsequently perform a RDN procedure

1) to verify the cutoff value (RNS-induced systolic BP change <20mmHg in post-RDN patients) could be a useful clinical endpoint in RDN therapy.

Hypotheses:

We hypothesize that an RNS-induced SBP increase of <20 mmHg in bilateral proximal main renal arteries immediately after RDN was associated with significant BP reductions 6 months following RDN. RNS-induced SBP changes could predict RDN response and even guide RDN strategies

Study design: Investigator initiated, single center, prospective study Patient population: 60 patients (20 - 80 years old) Patients with HTN.

1) 24-hour ambulatory blood pressure monitoring (ABPM) was >130 or DBP >80 mmHg

Exclusion criteria:

1. Unsuitable renal artery anatomy (main renal artery lumen diameter ≤3 mm or a total length <20 mm of the main arteries).
2. Secondary hypertension, including hyperaldosteronism, pheochromocytoma, renal artery stenosis(>50% stenosis in one or both arteries)
3. Pregnancy

Intervention:

RNS-guided RDN will be performed

1. Group A (N=35): RNS-induced SBP increase of <20 mmHg in bilateral proximal main renal arteries immediately after RDN
2. Group B(N=25): RNS-induced SBP increase of >20 mmHg in bilateral proximal main renal arteries immediately after RDN Then we will further divided Group B into Group C (N=8): observation group Group D(N=17): intensive intervention group (intensive -RDN again and the goal was post RNS-induced SBP change <20 mmHg)

Primary end-points:

The primary end points were the low RNS-induced systolic BP changes after RDN, was associated with the lower 24-hour SBP.

ELIGIBILITY:
Inclusion Criteria:

Patients with hypertension (HTN), including

1. 24-hour ambulatory blood pressure >130/ 80 mmHg
2. Age 20-80 years
3. Glomerular filtration rate >45 mL/min

Exclusion Criteria:

1. Unsuitable renal artery anatomy computed tomographic angiography (main renal artery lumen diameter ≤3 mm or a total length <20 mm of the main arteries).
2. untreated secondary HTN, including hyperaldosteronism, pheochromocytoma, renal artery stenosis(>50% stenosis)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-24 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
arterial blood pressure response | during procedure
  Main study parameter will be the arterial blood pressure response to RNS immediately after RDN.

SECONDARY OUTCOMES:
blood pressure at 6 months | 6 months after the intervention
  24 hours Blood pressure at 6 months after the intervention
blood pressure at 12 months | 12 months after the intervention
  24 hours Blood pressure at 12 months after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Rodeheffer RJ. Hypertension and heart failure: the ALLHAT imperative. Circulation. 2011 Oct 25;124(17):1803-5. doi: 10.1161/CIRCULATIONAHA.111.059303. No abstract available. PMID 22025634
- [Background] Bhatt DL, Kandzari DE, O'Neill WW, D'Agostino R, Flack JM, Katzen BT, Leon MB, Liu M, Mauri L, Negoita M, Cohen SA, Oparil S, Rocha-Singh K, Townsend RR, Bakris GL; SYMPLICITY HTN-3 Investigators. A controlled trial of renal denervation for resistant hypertension. N Engl J Med. 2014 Apr 10;370(15):1393-401. doi: 10.1056/NEJMoa1402670. Epub 2014 Mar 29. PMID 24678939
- [Background] Townsend RR, Mahfoud F, Kandzari DE, Kario K, Pocock S, Weber MA, Ewen S, Tsioufis K, Tousoulis D, Sharp ASP, Watkinson AF, Schmieder RE, Schmid A, Choi JW, East C, Walton A, Hopper I, Cohen DL, Wilensky R, Lee DP, Ma A, Devireddy CM, Lea JP, Lurz PC, Fengler K, Davies J, Chapman N, Cohen SA, DeBruin V, Fahy M, Jones DE, Rothman M, Bohm M; SPYRAL HTN-OFF MED trial investigators*. Catheter-based renal denervation in patients with uncontrolled hypertension in the absence of antihypertensive medications (SPYRAL HTN-OFF MED): a randomised, sham-controlled, proof-of-concept trial. Lancet. 2017 Nov 11;390(10108):2160-2170. doi: 10.1016/S0140-6736(17)32281-X. Epub 2017 Aug 28. PMID 28859944
- [Background] Kandzari DE, Bohm M, Mahfoud F, Townsend RR, Weber MA, Pocock S, Tsioufis K, Tousoulis D, Choi JW, East C, Brar S, Cohen SA, Fahy M, Pilcher G, Kario K; SPYRAL HTN-ON MED Trial Investigators. Effect of renal denervation on blood pressure in the presence of antihypertensive drugs: 6-month efficacy and safety results from the SPYRAL HTN-ON MED proof-of-concept randomised trial. Lancet. 2018 Jun 9;391(10137):2346-2355. doi: 10.1016/S0140-6736(18)30951-6. Epub 2018 May 23. PMID 29803589
- [Background] Azizi M, Schmieder RE, Mahfoud F, Weber MA, Daemen J, Davies J, Basile J, Kirtane AJ, Wang Y, Lobo MD, Saxena M, Feyz L, Rader F, Lurz P, Sayer J, Sapoval M, Levy T, Sanghvi K, Abraham J, Sharp ASP, Fisher NDL, Bloch MJ, Reeve-Stoffer H, Coleman L, Mullin C, Mauri L; RADIANCE-HTN Investigators. Endovascular ultrasound renal denervation to treat hypertension (RADIANCE-HTN SOLO): a multicentre, international, single-blind, randomised, sham-controlled trial. Lancet. 2018 Jun 9;391(10137):2335-2345. doi: 10.1016/S0140-6736(18)31082-1. Epub 2018 May 23. PMID 29803590
- [Background] Bohm M, Mahfoud F, Townsend RR, Kandzari DE, Pocock S, Ukena C, Weber MA, Hoshide S, Patel M, Tyson CC, Weil J, Agdirlioglu T, Fahy M, Kario K. Ambulatory heart rate reduction after catheter-based renal denervation in hypertensive patients not receiving anti-hypertensive medications: data from SPYRAL HTN-OFF MED, a randomized, sham-controlled, proof-of-concept trial. Eur Heart J. 2019 Mar 1;40(9):743-751. doi: 10.1093/eurheartj/ehy871. PMID 30608521
- [Background] Liu H, Chen W, Lai Y, Du H, Wang Z, Xu Y, Ling Z, Fan J, Xiao P, Zhang B, Wang J, Gyawali L, Zrenner B, Woo K, Yin Y. Selective Renal Denervation Guided by Renal Nerve Stimulation in Canine. Hypertension. 2019 Sep;74(3):536-545. doi: 10.1161/HYPERTENSIONAHA.119.12680. Epub 2019 Jul 22. PMID 31327262
- [Background] Gal P, de Jong MR, Smit JJ, Adiyaman A, Staessen JA, Elvan A. Blood pressure response to renal nerve stimulation in patients undergoing renal denervation: a feasibility study. J Hum Hypertens. 2015 May;29(5):292-5. doi: 10.1038/jhh.2014.91. Epub 2014 Oct 23. PMID 25339295